CLINICAL TRIAL: NCT01756885
Title: Extended Duration Varenicline for Smoking Among Cancer Patients: A Clinical Trial
Brief Title: Extended Varenicline Treatment for Smoking Among Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01CA165001 (NIH); NCT02851901 (obsolete NCT alias)
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Nicotine Dependence
Keywords: Smoking cessation; Nicotine dependence; Varenicline; Chantix; Cancer
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Neoplasms | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Varenicline Treatment (Active Comparator): 12 weeks of active varenicline + 12 weeks of placebo + smoking cessation counseling
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Days 85-168: Placebo - 1.0mg twice daily orally
  Interventions: Drug: Varenicline; Drug: Placebo; Behavioral: Smoking Cessation Counseling
- Extended Varenicline Treatment (Experimental): 24 weeks of active varenicline + smoking cessation counseling
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-168: 1.0mg twice daily orally
  Interventions: Drug: Varenicline; Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Drug: Varenicline — Varenicline was used in accordance with FDA approved labeling: Day 1-Day 3 (0.5mg once daily); Day 4-Day 7 (0.5mg twice daily); and Day 8-Day 84 (1.0mg twice daily).
  Other Names: Chantix
Drug: Placebo — On Day 85, participants randomized to standard therapy will be given placebo pills (resembling the 1.0mg pills),
  Arms: Standard Varenicline Treatment
Behavioral: Smoking Cessation Counseling — Behavioral Counseling (from Week 0 - Week 18)
  The counseling protocol was based on PHS guidelines for smoking cessation treatment (Fiore et al., 2008), used in our past studies with cancer patients (Schnoll et al., 2010a) and in our ongoing cessation trial at NU (R01 DA025078). Counseling is included given its efficacy at helping smokers quit (Fiore et al., 2008) and to increase study retention. Counseling is provided to both treatment arms through Week 18 to equate for time and attention across arms and since this method was used in varenicline clinical trials (Gonzales et al., 2006) and in our extended therapy trial (Schnoll et al., 2010b). In-person counseling was selected for most sessions to ensure adequate monitoring of participant safety and adherence throughout the trial.

SUMMARY:
Upwards of 33-50% of cancer patients who smoked prior to diagnosis continue to smoke following diagnosis and treatment. With medical advances in cancer care yielding a growing constituency of cancer survivors, addressing nicotine dependence in this population is a priority. While PHS guidelines recommend acute treatment durations with approved medications for tobacco use, extending the duration of treatment beyond the standard treatment duration significantly increases quit rates, reduces the risk for a relapse, and promotes recovery to abstinence following a lapse. Varenicline may be particularly effective for cancer patients given the drug's beneficial effects on affect and cognition. In this trial, 374 cancer patients will be randomized to standard varenicline treatment (12 weeks active + 12 weeks placebo) or extended varenicline treatment (24 weeks active). The investigators hypothesize that 1) Extended varenicline therapy will increase 24- and 52-week biochemically-confirmed abstinence versus standard varenicline treatment, 2) Quality of life will be rated higher in the extended therapy group versus the standard therapy group, and there will be no significant differences between groups in terms of severe side effects, and 3) Improved affect and reduced cognitive impairment will mediate the effect of extended therapy on quit rates.

DETAILED DESCRIPTION:
BACKGROUND

Prevalence of Smoking among Cancer Patients

The rate of smoking among individuals with cancer who are age 40 or under are substantially higher (38-40%) than rates of smoking in the comparable age group in the general population (~26%; Bellizzi et al., 2005; Coups & Ostroff, 2005). Studies with patients that have traditional tobacco-related cancers show extremely high rates of smoking; upwards of 50% of head and neck (Duffy et al., 2008) and lung (Cooley et al., 2009) cancer patients report current smoking. However, high rates of smoking are not unique to such traditional tobacco-related disease sites. Significant rates of current smoking have been reported among testicular (19%; Shinn et al., 2007), prostate (16-17%; Gong et al., 2008; Pantarotto et al., 2007), cervical (21%; Beesley et al., 2008), breast (19%; Li et al., 2009), bladder (18%; Blanchard et al., 2008), esophageal (39%; Sundelof et al., 2008), colorectal (22%; Vincenzi et al., 2009), and lymphoma (19%; Geyer et al., 2010) cancer patients. Overall, about one-third to one-half of cancer patients who were smokers prior to their diagnosis continue to smoke following diagnosis (Gritz et al., 2006).

Adverse Health Consequences of Smoking among Individuals with Cancer

Continued smoking by cancer patients has been associated with diminished QOL, reduced survival probability and duration, and increased risk for disease recurrence and a second primary tumor (Gritz et al., 2006; 2007). Continued smoking by cancer patients is associated with greater treatment side effects or diminished QOL among head and neck (Duffy et al., 2007; Zevallos et al., 2009), lung (Daniel et al., 2009), prostate (Ku et al., 2009), and a heterogeneous group of (Schnoll et al., 2010a) cancer patients. A recent meta-analysis of studies with lung cancer patients found that continued smoking was associated with an increased risk of death, recurrence, and a second primary tumor (Parsons et al., 2010). Likewise, studies with head and neck cancer patients have reported that patients who continue to smoke following their diagnosis have a lower survival rate and an increased risk for a recurrence and a second primary tumor (Browman et al., 2002; Hilgert et al., 2009; Fortin et al., 2009; Leon et al., 2009). Continued smoking has also been associated with reduced survival among breast (Aksoy et al., 2007), lymphoma (Geyer et al., 2010), esophageal (Sundelof et al., 2008), prostate (Gong et al., 2008), cervical (Coker et al., 2009), and bladder (Aveyard et al., 2002) cancer patients and with an increased risk of recurrence or a second primary tumor among bladder (Fleshner et al., 1999), breast (Li et al., 2009), lymphoma (Moser et al., 2006), and colorectal (Jacobson et al., 1994) cancer patients. Continued smoking may worsen prognosis by reducing the effectiveness of chemotherapy (Duarte et al., 2008; van der Bol et al., 2007; Vincenzi et al., 2009; Hotta et al., 2008) and radiotherapy (Browman et al., 1993).

Nicotine Dependence Treatments for Those with Cancer

Very few smoking cessation trials have been conducted with this population (Gritz et al., 2006; 2007) and many of these past trials have used small samples and relied on self-report for smoking abstinence outcomes (de Moor et al., 2008). After nearly two decades of research in this area, not a single smoking cessation randomized clinical trial has yielded significant treatment effects (excluding Emmons et al., 2009, which studied adult survivors of childhood cancer; de Moor et al., 2008). Nurse-led (Griebel et al., 1998; Stanislaw & Wewers, 1994; Wewers et al., 1994), physician-led (Browning et al., 2000; Gritz et al., 1993; Schnoll et al., 2003b), and behavioral (Schnoll et al., 2005; Wakefield et al., 2004) smoking cessation trials have failed to yield treatment effects for cancer patients. Our recent clinical trial with bupropion (Schnoll et al., 2010a) found no main effect for the medication, but bupropion increased abstinence rates, reduced withdrawal symptoms, and improved QOL more for patients with depression, vs. those without depression. Lastly, a very recent varenicline study reported end-of-treatment quit rates of 34%, vs. 14% for the comparison group (OR = 3.14), and a side effect profile that mirrored the general population (Park et al., 2011). While these data are encouraging, as were reported feasibility data, the study was under-powered (n = 49) and did not use a randomized design. Thus, there is currently no empirically-based treatment model for addressing nicotine dependence in the oncologic context. As such, a recent NCI meeting, with representatives from NCI cancer centers, concluded that the evaluation of novel smoking cessation interventions for cancer patients is a critical priority (Morgan et al., 2010).

A Novel Treatment for Cancer Patients who Smoke: Extended Duration Varenicline Thus, nicotine dependence treatments for cancer patients may show greater efficacy if they adequately address the patient's relatively high level of nicotine dependence, risk for psychological distress and cognitive impairment, and delayed relapse process. We hypothesize that extended duration varenicline (24-weeks) will address these barriers to cessation and significantly increase quit rates, vs. standard varenicline treatment (12 weeks).

Our rationale for selecting varenicline is as follows. First, the high rate of nicotine dependence among cancer patients underscores the need to include a pharmacotherapy as part of treatment. Varenicline is currently the most efficacious FDA-approved medication for nicotine dependence, yielding quit rates that significantly exceed those produced by bupropion (Gonzales et al., 2006; Jorenby et al., 2006) and nicotine patch (Aubin et al., 2008; Biazzo et al., 2010; Stapleton et al., 2008). Second, varenicline mitigates adverse psychological effects and cognitive impairment associated with quitting smoking (Patterson et al., 2009; Smith et al., 2009; Philip et al., 2009; Rollema et al., 2009; Sofuoglu et al., 2009). The anti-depressant-like (Rollema et al., 2009) and cognitive enhancing (Loughead et al., 2010) effects of varenicline is consistent with what we know about how varenicline works. As a nicotinic acetylcholine receptor (nAChRs) partial agonist, varenicline binds to nAChRs and blocks the entry of nicotine (from smoking) into the receptor and stimulates a moderate release of dopamine. This reduces the rewarding effects of smoking and reduces withdrawal symptoms (Rollema et al., 2009). Preclinical studies also indicate that α4β2 nAChRs subtypes are critical for cognition (Levin et al., 2006) and stimulation of these receptors by varenicline yields improved cognitive function (Loughead et al., 2010). Likewise, animal studies indicate that the simultaneous activation and desensitization of nAChRs receptors produced by nicotinic partial agonists like varenicline can yield antidepressant-like effects (Mineur & Picciotto, 2010), which underlies current evaluations of varenicline as a treatment for major depression. Third, varenicline is efficacious and safe for treating nicotine dependence among various clinical populations, including: cardiovascular disease patients (Rigotti et al., 2010), COPD patients (Tashkin et al., 2010), smokers with comorbid alcohol (Hays et al., 2010) and cocaine (Poling et al., 2010) dependence, and smokers with comorbid affective or psychotic disorders (McClure et al., 2010; Smith et al., 2009; Philip et al., 2009). It has been shown to be safe when taken over 52 weeks (Williams et al., 2007). Although there have been reports of adverse psychiatric events following varenicline use, leading the FDA to mandate a boxed warning for varenicline, pooled data from controlled efficacy trials (Cahill et al., 2009; Tonstad et al., 2010), effectiveness trials (McClure et al., 2010), and large cohort studies (Gunnell et al., 2009; Kasliwal et al., 2009) demonstrate that varenicline is safe for treating nicotine dependence, even among smokers with psychiatric comorbidity, including depression (Stapleton et al., 2008; McClure et al., 2010; Steinberg et al., 2010).

Our rationale for selecting an extended duration treatment is as follows. First, we have shown, in a placebo-controlled randomized trial with general population smokers, that 24-weeks of transdermal nicotine, vs. the standard 8-weeks, increases 6-month quit rates by an OR of 1.81 (32% vs. 20%; Schnoll et al., 2010b). Second, and importantly, extending treatment with the nicotine patch to 24-weeks significantly helps smokers with high levels of nicotine dependence and cognitive impairment, in particular, to overcome their liability to relapse (see below). While extended therapy with transdermal nicotine did not offset the effect of depression symptoms on relapse rates, the quit rate among depressed smokers in extended treatment was almost 2-times higher than it was for depressed smokers in standard treatment (see below). Third, we showed in our placebo-controlled randomized clinical trial with general population smokers (Schnoll et al., 2010b) that extending treatment with transdermal nicotine to 24-weeks (vs. 8-weeks) significantly reduced the probability that smokers would experience a lapse and, importantly, increased the likelihood that smokers would recover to abstinence following a lapse. Extended duration treatment offered smokers who lapsed the opportunity to re-start their quit attempt and eventually achieve abstinence. Thus, extended duration varenicline may be particularly efficacious at addressing the barriers to cessation that are evident among cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older who self-report smoking at least 5 cigarettes (menthol and non-menthol) per day, on average, for the last 6 months.
2. Current cancer diagnosis (all sites) or diagnosis within the past 5 years.
3. Karnofsky Score of >50 or ECOG Performance Status score of <2 within 6 months of enrollment.
4. Able to use varenicline safely, based on a medical evaluation including medical history and physical examination, and psychiatric evaluation.
5. Residing in the geographic area for at least 12 months.
6. Women of childbearing potential (based on medical history and physical exam) must consent to use a medically accepted method of birth control (e.g., condoms and spermicide, oral contraceptive, Depo-Provera injection, contraceptive patch, tubal ligation) or abstain from sexual intercourse during the time they are taking study medication and for at least one month after the medication period ends.
7. Able to communicate fluently in English.
8. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent/HIPAA form.

Exclusion Criteria:

Smoking Behavior

1. Current enrollment or plans to enroll in another smoking cessation program in the next 12 months.
2. Regular (daily) use of chewing tobacco, snuff, snus, cigars, cigarillos, or pipes.
3. Current use or plans to use nicotine substitutes (gum, patch, lozenge, e-cigarette) or smoking cessation treatments in the next 12 months.

   1. Note: Once participants are found eligible for the study, they are told they should refrain from using any nicotine replacement therapy (NRT) for the duration of the study. If a subject reports an isolated (non-daily) instance of NRT use during the study, they may be permitted to continue.

Alcohol/Drug Exclusion Criteria

1. Diagnosis of substance abuse or dependence that has been unstable in the past year.
2. Positive urine drug screen (for cocaine, opioids, or methamphetamines) at the Intake Session (unless taking opiate for pain management).
3. Breath Alcohol Concentration (BrAC) assessment greater than or equal to 0.01 at the Intake Session.
4. Current alcohol consumption that exceeds 25 standard alcoholic drinks/week.

Medication Exclusion Criteria

Current use or recent discontinuation (within last 14 days) of the following medications:

1. Other smoking cessation medications (e.g. Zyban, Wellbutrin, Wellbutrin SR, Chantix)

   a. Note: Once participants are found eligible for the study, they are instructed to only use the smoking cessation medication provided to them by the study staff. If a subject reports an isolated (non-daily) instance of using a non-study smoking cessation medication, the study physician and PI will evaluate the situation and determine if it is safe for the subject to continue participation.
2. Anti-psychotic medications.
3. Bipolar Disorder medications.

Medical Exclusion Criteria

1. Women who are pregnant, planning a pregnancy within the next 12 months, or lactating.
2. History of epilepsy or seizure disorder (history of seizure requires Study Physician approval).
3. History of kidney disease, including transplant.
4. Uncontrolled hypertension (SBP >160 or DBP >100).

   a. Note: If a participant presents with blood pressure greater than 160/100 at sessions occurring on Week 0 (Pre-Quit) or at any other point during the treatment period, they will not be provided with/able to continue on medication unless the study physician grants approval.
5. History of heart disease, stroke or MI, unstable angina, abnormal heart rhythms, or tachycardia (if stable, requires Study Physician approval).
6. Abnormal ECG (unless approved by Study Physician).
7. Any suicide risk score on MINI, current suicidal ideation on Columbia scale, or self-reported suicide attempt.
8. Current or past diagnosis of psychotic or bipolar disorder, as determined by self-report & MINI.
9. Current diagnosis of unstable and untreated major depression, as determined by self-report & MINI (eligible if stable for >30 days).
10. Previous allergic reaction to varenicline.

General Exclusion Criteria

1. Any medical condition or concomitant medication that could compromise subject safety or treatment, as determined by the Principal Investigator and/or Study Physician.
2. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2013-01; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Schnoll, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Varenicline Treatment: 12 weeks of active varenicline + 12 weeks of placebo + smoking cessation counseling
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-84: 1.0mg twice daily orally
  Days 85-168: Placebo - 1.0mg twice daily orally
  Varenicline
  Placebo
  Smoking Cessation Counseling
- Extended Varenicline Treatment: 24 weeks of active varenicline + smoking cessation counseling
  Day 1-3: 0.5mg once daily orally Day 4-7: 0.5mg twice daily orally Day 8-168: 1.0mg twice daily orally
  Varenicline
  Smoking Cessation Counseling
Period: Overall Study
Arm/Group | Standard Varenicline Treatment | Extended Varenicline Treatment
Started | 102 | 105
Completed | 79 | 79
Not Completed | 23 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Varenicline Treatment | Extended Varenicline Treatment | Total
Number analyzed (Participants) | 102 | 105 | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 81 | 163
  >=65 years | 20 | 24 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.5) | 58.00 (9.4) | 58.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 59 | 105
  Male | 56 | 46 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 96 | 100 | 196
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 31 | 57
  White | 72 | 72 | 144
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 102 | 105 | 207
Fagerström Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Scale range from 0-10. Higher score indicates greater nicotine dependence.
  units on a scale | 4.6 (2.2) | 4.4 (2.1) | 4.5 (2.1)
Karnofsky Performance Score [Mean (Standard Deviation); unit: units on a scale] — The Karnofsky Performance Scale is an assessment tool for functional impairment. Scale range from 0-100. Higher score indicates less functional impairment.
  units on a scale | 91.7 (11.7) | 92.1 (10.9) | 91.9 (11.2)
ECOG Performance Status [Mean (Standard Deviation); unit: units on a scale] — The ECOG Performance Scale is used to assess how a patient's cancer is progressing and assess how the disease affects the daily living abilities of the patient. Scale range from 0-5. Higher score indicates further progression of cancer.
  units on a scale | 0.25 (0.43) | 0.25 (0.44) | 0.25 (0.43)
Breath carbon monoxide [Mean (Standard Deviation); unit: units on a scale] — Breath carbon monoxide is the level of carbon monoxide in a person's exhalation. The minimum score is 0, while there is no maximum score. Higher scores indicate a higher level of carbon monoxide in parts per million (ppm) in breath.
  units on a scale | 18.2 (11.3) | 19.7 (11.0) | 19.0 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: 7-day CO-verified Tobacco Abstinence
Description: Number of Participants with Verified 7 Day Tobacco Abstinence.
Time Frame: Weeks 24 & 52
Measure: Number; unit: participants
Arm/Group | Standard Varenicline Treatment | Extended Varenicline Treatment
Number analyzed (Participants) | 102 | 105
participants
  Week 24 | 28 | 32
  Week 52 | 16 | 17

2. Secondary Outcome: Quality of Life at Week 24 and 52
Description: The Short-Form Health Survey (SF-12) assesses Quality of Life (QOL). Scale range from 12 - 47. Higher score indicates worse quality of life.
Time Frame: Weeks 24 & 52
Population: Difference in number of participants at Weeks 24 and 52 are due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Varenicline Treatment | Extended Varenicline Treatment
Number analyzed (Participants) | 52 | 56
score on a scale
  Week 24 | 38.75 (6.17) | 38.46 (5.90)
  Week 52: number analyzed (Participants) | 51 | 47
  Week 52 | 38.06 (6.81) | 36.91 (6.30)

3. Other Pre Specified Outcome: Number of Participants With Continuous Abstinence
Description: No smoking from baseline to time-point, after a 2-week grace period.
Time Frame: Weeks 12, 24, and 52
Measure: Number; unit: participants
Arm/Group | Standard Varenicline Treatment | Extended Varenicline Treatment
Number analyzed (Participants) | 102 | 105
participants
  Week 24 | 19 | 22
  Week 52 | 11 | 16

ADVERSE EVENTS:
Time Frame: 53 weeks
Description: Research staff member completed side effect assessments and determined the severity of the adverse events; the relationship of the event to the study drug and the decision on the course of action for the participant was decided by the site physicians and psychologists after review of the report. Participants were monitored for the development of adverse events by assessing side effects at each assessment time-point, as well as through open-ended questions during assessments.
Arm/Group | Standard Varenicline Treatment | Extended Varenicline Treatment
All-Cause Mortality (participants affected / at risk) | 4/102 | 1/105
Serious Adverse Events (participants affected / at risk) | 9/102 | 13/105
Other Adverse Events (participants affected / at risk) | 27/102 | 25/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Varenicline Treatment (N=102) | Extended Varenicline Treatment (N=105)
Dehydration, fluid build-up (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dysphagia and difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Facial edema (General disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fever and swelling (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Confusion (General disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anxiety (panic) attack (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation and bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Second cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Radiation burn infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cracked ribs (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute kidney injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Injury from fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headaches (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 4 (4) | 1 (1)
Cancer progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blood loss (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Enterocolotis infection (Infections and infestations) | 1 (2) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Varenicline Treatment (N=102) | Extended Varenicline Treatment (N=105)
Weakness (General disorders) | 2 | 0
Skin swelling, rash, or redness (Skin and subcutaneous tissue disorders) | 3 | 1
Depression (Psychiatric disorders) | 21 | 20
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cancer recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Suicidality (Psychiatric disorders) | 2 | 0
Nausea, abdominal pain (Gastrointestinal disorders) | 6 | 4
Irritability (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Agitation (Psychiatric disorders) | 4 | 9
Hostility (Psychiatric disorders) | 1 | 7
High cholesterol (Blood and lymphatic system disorders) | 1 | 0
Hemorrhoids (Skin and subcutaneous tissue disorders) | 1 | 0
Heart attack (Cardiac disorders) | 0 | 1
Headache (General disorders) | 0 | 2
Dizziness (General disorders) | 3 | 1
Gout (worsening) (General disorders) | 1 | 0
Pins and needles feeling (General disorders) | 0 | 1
Fainting (General disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholecytstosis (Gastrointestinal disorders) | 1 | 0
Cirrhosis (Gastrointestinal disorders) | 1 | 0
Bracial plexopathy (Nervous system disorders) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hyperglycemia (Endocrine disorders) | 1 | 0
Arterial injury (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT01756885/Prot_SAP_000.pdf